CLINICAL TRIAL: NCT02261909
Title: New Prognostic Kidney Function Markers in Emergency Patients
Brief Title: New Prognostic Kidney Function Markers in Emergency Patients New Markers of Kidney Function in ED Patients
Status: Withdrawn | Type: Observational
Why Stopped: Study failed to receive final approvement
Sponsor: Krankenhaus Barmherzige Brüder, Regensburg (Other)
Collaborators: Astute Medical, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 1
Record Dates: First submitted 2014-10-03; First posted 2014-10-10 (Estimated); Last update posted 2022-08-22 (Actual); Status verified 2022-08

CONDITIONS: Acute Kidney Injury; Contrast Media
Keywords: Emergency Medicine; diagnosis
MeSH Terms: conditions — Acute Kidney Injury; Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum, urine
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- normal creatinine: pts receiving an iv-contrast enhanced CT with normal baseline renal function
- elevated creatinine: pts receiving an iv-contrast enhanced CT with abnormal baseline renal function

SUMMARY:
NephroCheck is measuring the concentration of a certain protein combination in the urine of patients. In elevated values there is a probability of renal failure (already proven in intensive care patients). The investigators would like to investigate whether the investigators can predict renal failure in patients receiving contrast enhanced CT's in the emergency department. That would lead to an earlier nephrologist consult in those patients.

DETAILED DESCRIPTION:
The use of contrast agents can - especially in already in impaired renal function - lead to a decline in real function. The contrast enhanced CT is especially in emergency patients an important diagnostic tool for example in the detection of pulmonary embolism or mesenteric ischemia. Creatinine has been used as a marker for real function so far. But the investigators all know that creatinine is not a perfect marker especially as it is influenced by age, sex, weight and muscle mass. Especially in the diagnosis of acute renal failure creatinine does not allow and recent change in the kidney function.

This prospective, unicentric study should therefore investigate two new markers in emergency patients who need an emergency contrast enhanced CT to early predict pending kidney function decline.

ELIGIBILITY:
Inclusion Criteria:

* patients in the emergency department who have the indication for contrast enhanced CT and a predicted hospital admission time of 48 hours or longer.

Exclusion Criteria:

* children, pregnant women
* dialysis
* patients with kidney transplants
* patients on steroids or further immunocompromised

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients in the in emergency department who have the indication for contrast enhanced CT and a predicted hospital admission time of 48 hours or longer.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2015-05; Primary Completion 2016-05 (Estimated); Study Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
Renal function | participants will be followed for the duration of hospital stay, an expected average of 7 days
  renal function at discharge from hospital (creatinine and BUN measured at day of discharge)

SECONDARY OUTCOMES:
Requirement for dialysis | participants will be followed for the duration of hospital stay, an expected average of 7 days
  dialysis required throughout hospital stay
Admission to ICU | participants will be followed for the duration of hospital stay, an expected average of 7 days
  admission to ICU required throughout hospital stay

CONTACTS AND LOCATIONS:
Overall Officials: Jan Braess, Prof, Study Chair — Krankenhaus Barmherzige Brüder
Locations (1):
- Krankenhaus Barmherzige Brueder, Regensburg, Bavaria, Germany

REFERENCES:
- [Background] Meersch M, Schmidt C, Van Aken H, Martens S, Rossaint J, Singbartl K, Gorlich D, Kellum JA, Zarbock A. Urinary TIMP-2 and IGFBP7 as early biomarkers of acute kidney injury and renal recovery following cardiac surgery. PLoS One. 2014 Mar 27;9(3):e93460. doi: 10.1371/journal.pone.0093460. eCollection 2014. PMID 24675717
- [Background] Olden M, Corre T, Hayward C, Toniolo D, Ulivi S, Gasparini P, Pistis G, Hwang SJ, Bergmann S, Campbell H, Cocca M, Gandin I, Girotto G, Glaudemans B, Hastie ND, Loffing J, Polasek O, Rampoldi L, Rudan I, Sala C, Traglia M, Vollenweider P, Vuckovic D, Youhanna S, Weber J, Wright AF, Kutalik Z, Bochud M, Fox CS, Devuyst O. Common variants in UMOD associate with urinary uromodulin levels: a meta-analysis. J Am Soc Nephrol. 2014 Aug;25(8):1869-82. doi: 10.1681/ASN.2013070781. Epub 2014 Feb 27. PMID 24578125
- [Background] Kellum JA, Lameire N; KDIGO AKI Guideline Work Group. Diagnosis, evaluation, and management of acute kidney injury: a KDIGO summary (Part 1). Crit Care. 2013 Feb 4;17(1):204. doi: 10.1186/cc11454. PMID 23394211
- [Background] Lameire N, Kellum JA; KDIGO AKI Guideline Work Group. Contrast-induced acute kidney injury and renal support for acute kidney injury: a KDIGO summary (Part 2). Crit Care. 2013 Feb 4;17(1):205. doi: 10.1186/cc11455. PMID 23394215
- [Background] Risch L, Lhotta K, Meier D, Medina-Escobar P, Nydegger UE, Risch M. The serum uromodulin level is associated with kidney function. Clin Chem Lab Med. 2014 Dec;52(12):1755-61. doi: 10.1515/cclm-2014-0505. PMID 24933630
- [Background] Bihorac A, Chawla LS, Shaw AD, Al-Khafaji A, Davison DL, Demuth GE, Fitzgerald R, Gong MN, Graham DD, Gunnerson K, Heung M, Jortani S, Kleerup E, Koyner JL, Krell K, Letourneau J, Lissauer M, Miner J, Nguyen HB, Ortega LM, Self WH, Sellman R, Shi J, Straseski J, Szalados JE, Wilber ST, Walker MG, Wilson J, Wunderink R, Zimmerman J, Kellum JA. Validation of cell-cycle arrest biomarkers for acute kidney injury using clinical adjudication. Am J Respir Crit Care Med. 2014 Apr 15;189(8):932-9. doi: 10.1164/rccm.201401-0077OC. PMID 24559465
- [Background] Kashani K, Al-Khafaji A, Ardiles T, Artigas A, Bagshaw SM, Bell M, Bihorac A, Birkhahn R, Cely CM, Chawla LS, Davison DL, Feldkamp T, Forni LG, Gong MN, Gunnerson KJ, Haase M, Hackett J, Honore PM, Hoste EA, Joannes-Boyau O, Joannidis M, Kim P, Koyner JL, Laskowitz DT, Lissauer ME, Marx G, McCullough PA, Mullaney S, Ostermann M, Rimmele T, Shapiro NI, Shaw AD, Shi J, Sprague AM, Vincent JL, Vinsonneau C, Wagner L, Walker MG, Wilkerson RG, Zacharowski K, Kellum JA. Discovery and validation of cell cycle arrest biomarkers in human acute kidney injury. Crit Care. 2013 Feb 6;17(1):R25. doi: 10.1186/cc12503. PMID 23388612